CLINICAL TRIAL: NCT02969109
Title: Clinical Validation of a Urine-based Assay With Genomic and Epigenomic Markers for Predicting Recurrence During Surveillance for Non-muscle Invasive Bladder Cancer
Brief Title: Validation of a Urine-based Assay With Genomic Markers for Predicting Recurrence for Non-muscle Invasive Bladder Cancer
Status: Completed | Type: Observational
Sponsor: Genomic Health®, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 14-006
Record Dates: First submitted 2016-11-14; First posted 2016-11-21 (Estimated); Last update posted 2021-03-02 (Actual); Status verified 2021-02

CONDITIONS: Non-muscle Invasive Bladder Cancer
MeSH Terms: conditions — Non-Muscle Invasive Bladder Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine and tissue
Oversight: Data Monitoring Committee: No

SUMMARY:
A study to validate, in a prospective manner, the ability of the predefined Genomic Health bladder cancer assay to detect recurrence in patients undergoing surveillance for non-muscle invasive bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

* Patients with a prior diagnosis of non-muscle invasive, ≤T1, urothelial cell carcinoma of the bladder scheduled to undergo surveillance cystoscopy.

Exclusion Criteria:

* Patients younger than 18 years
* Patients with a diagnosis of small cell carcinoma, adenocarcinoma or squamous cell carcinoma of the bladder
* Patients who have had a cystectomy or prior diagnosis of muscle invasive disease (T2 or greater)
* Patients who are unable or unwilling to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Non-muscle invasive bladder cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 417 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2018-09-18 (Actual); Study Completion 2018-09-18 (Actual)

PRIMARY OUTCOMES:
The recurrence status based on the pathology results | 1 year
The Genomic Health bladder cancer assay results. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Institute for Prostate and Urologic Cancers - University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No